CLINICAL TRIAL: NCT01986985
Title: Comparison of 18F FDG PET/CT TO PET MRI
Acronym: PET/MR US
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 114-2013-GES-0014
Record Dates: First submitted 2013-11-06; First posted 2013-11-19 (Estimated); Results first posted 2015-05-04 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-02

CONDITIONS: Any Condition With a Clinical Indication for PET/CT Exam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm PET MRI (Other): single group evaluation of PET/MRI system scan for diagnostic quality of image
  Interventions: Device: PET/MRI system

INTERVENTIONS:
Device: PET/MRI system — Compared to PET CT
  Other Names: PET/MRI system inlcudes:; 3T MR750w Magnet; MR750w XRMw Gradient; PET/MRI Body Coil; Photon Detection Ring and PET Detectors; PET/MR Patient Table; PET Electronics (mounted to magnet) and Cables

SUMMARY:
The objective of this study is to gather image and associated data to of a pre-market PET/MRI scanner and to use the data for regulatory submission and future product development and marketing. Clinical data is required in order to test the MR attenuation correction of PET data. These aims can only be accomplished through a clinical study.

ELIGIBILITY:
Inclusion criteria

1. Subject must have a clinical indication for a PET/CT exam
2. Subject must be at least eighteen (18) years of age
3. Female subjects that are determined to be non-pregnant by a physician investigator or are demonstrated non-pregnant by negative urine pregnancy test administered within the 24 hour period before PET/CT imaging
4. Subject must be able to hear and understand instructions without assistive devices
5. Subject must provide written informed consent
6. Subject has the necessary mental capacity to understand instructions, and is able to comply with protocol requirements
7. Subject is able to remain still for duration of imaging procedure (approximately 60 minutes total for PET/MRI); and
8. Subject must be able to participate in a PET/MR imaging session within 1 hour of concluding their PET/CT exam.

Exclusion criteria

1. Subjects who have any axial diameter larger than 55 cm
2. Subjects with a weight greater than 499 lbs
3. Subjects that have metallic/conductive or electrically/magnetically active implants without MR Safe or MR Conditional labeling, with the exception of dental devices/fillings, surgical clips, and surgical staples determined to be safe for MRI scanning by a physician investigator
4. Subjects that have implants with MR Unsafe labeling;
5. Subjects that have implants labeled as MR Conditional by the manufacturer for which the allowable conditions are not expected to be achieved by the MR/PET environment or scan protocol;
6. Subjects who have a contraindication to MRI per the screening policy of the participating site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2014-01; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roee Lazebnik, MD, Study Director — GE Healthcare
Locations (2):
- United States (2):
  - University of California - San Francisco, San Francisco, California
  - Stanford University, Stanford, California

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm PET MRI: single group evaluation of PET/ MR for diagnostic quality of image
  PET/MRI system: Compared to PET CT
Period: Overall Study
Arm/Group | Single Arm PET MRI
Started | 58
Completed | 51
Not Completed | 7
Not completed — Withdrawal by Subject | 4
Not completed — Scan not completed due to malfunction | 3

BASELINE CHARACTERISTICS:
Population: Intent to treat
Arm/Group | Single Arm PET MRI
Number analyzed (Participants) | 58
Age, Customized [Number; unit: participants]
  Adult (>=18 years) | 58
Sex/Gender, Customized [Number; unit: participants]
  Male | 29
  Female | 29

OUTCOME MEASURES:

1. Primary Outcome: PET/MR Images Clinical Usefulness
Description: Clinically relevant images are obtained
Time Frame: 1 day
Population: Subjects with images successfully collected using PET/ MR
Measure: Number; unit: Participants
Arm/Group | Single Arm PET MRI
Number analyzed (Participants) | 58
Participants | 51

ADVERSE EVENTS:
Arm/Group | Single Arm PET MRI
Serious Adverse Events (participants affected / at risk) | 0/58
Other Adverse Events (participants affected / at risk) | 5/58
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm PET MRI (N=58)
Localized Warming (Skin and subcutaneous tissue disorders) | 4 (4)
Unilateral superficial skin injury of ear from head coil placement (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days